CLINICAL TRIAL: NCT05174026
Title: A Pilot Study on the Efficacy of Advanced 18F-FDG PET-MRI in Spine Stereotactic Radiosurgery
Brief Title: 18F-FDG PET-MRI for Planning and Follow-Up of Patients With Spine Tumors Treated With Spine Stereotactic Radiosurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-0788; NCI-2019-08261 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0788 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-09-10; First posted 2021-12-30 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Metastatic Malignant Neoplasm; Metastatic Malignant Neoplasm in the Bone
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (18F-FDG PET-MRI) (Experimental): Patients receive fludeoxyglucose F-18 IV over 1 minute, and then undergo PET-MRI over 1 hour, 30 days before radiation therapy, and 3 and 6 months after radiation therapy.
  Interventions: Other: Fludeoxyglucose F-18; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Other: Fludeoxyglucose F-18 — Given IV
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Procedure: Magnetic Resonance Imaging — Undergo 18F-FDG PET-MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo 18F-FDG PET-MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This trial studies how well 18F-FDG PET-MRI works for treatment planning in patients with spine tumors. Diagnostic procedures, such as 18F-FDG PET-MRI may help radiation oncologists plan the best treatment for spine tumors, as well as help in follow-up after radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the therapeutic efficacy of fludeoxyglucose F-18 (18F-FDG) positron emission tomography (PET)-magnetic resonance imaging (MRI) in spine stereotactic radiosurgery (SSRS) treatment planning compared to advanced MRI (aMRI) and conventional MRI (cMRI).

II. Determine the diagnostic accuracy of 18F-FDG PET-MRI in follow-up of patients treated with SSRS.

SECONDARY OBJECTIVES:

I. Analysis of the subset of patients who eventually suffer local treatment failure to determine patterns of failure and potential predictive PET/MRI features at baseline.

II. Analysis of the subset of patients who suffer complications of SSRS (e.g., vertebral compression fracture) to determine potential predictive imaging features.

OUTLINE:

Patients receive fludeoxyglucose F-18 intravenously (IV) over 1 minute, and then undergo PET-MRI over 1 hour, 30 days before radiation therapy, and 3 and 6 months after radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Consent to imaging study
* Presence of at least 1 lumbar vertebral body bone metastasis > 1 cm in shortest diameter and smaller than 75% of the vertebral body cross sectional area. Metastasis may be determined by pathology, or imaging appearance.
* Eligibility to receive SSRS (determined by treating radiation oncologists)
* Plan for single-fraction SSRS
* Standard-of-care spine MRI within 8 weeks of radiation therapy
* Ability to understand and willingness to sign a written informed consent document
* Non-English speaking participants will be included. Verbal Translation Preparative Sheet (VTPS) short form will be utilized in consenting non-English speaking participants.

Exclusion Criteria:

* Absolute or relative contra-indication to MRI, including presence of a pacemaker that requires involvement of cardiology/anesthesiology during the scan
* Prior directed radiation to the involved segment
* Contra-indication to gadolinium based contrast agents (e.g., allergy, pregnancy)
* Individuals younger than 18 years
* Hardware at the treatment level or hardware affecting visualization of the involved level on MRI
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Determine the therapeutic efficacy of fludeoxyglucose F-18 (18F-FDG) positron emission tomography (PET)-magnetic resonance imaging (MRI). | up to 6 months
Determine the diagnostic accuracy of 18F-FDG PET-MRI in follow-up of patients. | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Behrang Amini, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org